CLINICAL TRIAL: NCT03331432
Title: Targeting Endoplasmic Reticulum Stress to Correct Vascular Insulin Resistance and Glycemic Dysregulation
Brief Title: Effects of Dietary Supplement Tauroursodeoxycholic Acid on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jaume Padilla, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1203573
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ursodoxicoltaurine

STUDY DESIGN:
Intervention Model Description: Single-blinded randomized crossover study
Who Masked: Participant
Masking Description: Participants are not told which are placebo or tauroursodeoxycholic acid capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Taking daily placebo capsules for 4 weeks
  Interventions: Dietary Supplement: Placebo
- Tauroursodeoxycholic acid (Experimental): Taking tauroursodeoxycholic acid (1750 mg/day) capsules for 4 weeks
  Interventions: Dietary Supplement: Tauroursodeoxycholic acid

INTERVENTIONS:
Dietary Supplement: Tauroursodeoxycholic acid — Taking tauroursodeoxycholic acid (1750 mg/day) capsules for 4 weeks.
  Arms: Tauroursodeoxycholic acid
Dietary Supplement: Placebo — Taking daily placebo capsules for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of the present study is to determine if use of dietary supplement tauroursodeoxycholic acid enhances insulin-stimulated leg blood flow and glucose disposal.

DETAILED DESCRIPTION:
The notion that cellular stress lowers insulin-induced vasodilation is largely founded on ex vivo studies and experiments in rodents. However, it remains unknown if maintenance of cellular function with the use of dietary supplement tauroursodeoxycholic acid enhances vascular function in humans. The investigators test the hypothesis that daily administration of this dietary supplement enhances vascular function, particularly, insulin-stimulated leg blood flow and glucose disposal.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed by primary physician
* Body mass index less then 43 kg/m2

Exclusion Criteria:

* Recent weight gain or loss (>5% body weight in the last 3 months)
* Pregnancy
* Consumption of >14 alcoholic beverages per week
* Changes in the medication use or dose within the last 3 months
* Known cardiovascular or pulmonary disease
* Taking medication for advanced retinopathy or neuropathy
* Taking prescription anticoagulants
* Nicotine use

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Blood flow | Once at 4 weeks after the start of placebo and once at 4 weeks after the start of tauroursodeoxycholic acid
  Blood flow response during insulin clamp
Vascular function | Once at 4 weeks after the start of placebo and once at 4 weeks after the start of tauroursodeoxycholic acid
  Flow-mediated dilation
Insulin resistance | Once at 4 weeks after the start of placebo and once at 4 weeks after the start of tauroursodeoxycholic acid
  Glucose disposal rate during insulin clamp
Glucose tolerance | Once at 4 weeks after the start of placebo and once at 4 weeks after the start of tauroursodeoxycholic acid
  Glucose response to an oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Padilla, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No